CLINICAL TRIAL: NCT01178307
Title: Symptom Burden in Patients With Gastrointestinal Stromal Tumors (GISTs)
Brief Title: Symptom Inventory for Gastrointestinal Stromal Tumors
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Other Study IDs: 2010-0267
Record Dates: First submitted 2010-08-06; First posted 2010-08-10 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: GI cancers; GIST; Symptom Severity; Quality of Life; Questionnaire; M.D. Anderson Symptom Inventory; MDASI-GIST; patient-reported outcomes
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — Surveys and Questionnaires; Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Part 1: Patient interview and developmental questionnaires
  Interventions: Behavioral: Questionnaires; Behavioral: Interview
- Part 2: Content Expert Panel (doctors, nurses) + Patients and Caregivers Questionnaire Development
  Interventions: Behavioral: Questionnaires
- Part 3: Patient MDASI-GIST Questionnaire
  Interventions: Behavioral: MDASI-GIST Questionnaire

INTERVENTIONS:
Behavioral: Questionnaires — 10 minutes to complete 3 questionnaires for development of MDASI-GIST
  Other Names: survey
  Groups: Part 1; Part 2
Behavioral: Interview — Each interview will take approximately 30 minutes.
  Groups: Part 1
Behavioral: MDASI-GIST Questionnaire — Every 4 weeks for one year
  Other Names: survey
  Groups: Part 3

SUMMARY:
The goal of this research study is to better understand the symptoms experienced by patients with GIST.

There are 3 parts to this study. In Part 1, participants will complete 1 set of interviews and questionnaires about GIST symptoms. In Part 2, the importance of some symptoms to patients with GIST will be rated by doctors, nurses, patients, and family caregivers. In Part 3, participants will complete questionnaires about GIST symptoms over 1 year.

You are being asked to take part in Part 3 of the study.

DETAILED DESCRIPTION:
Symptom Questionnaires:

If you agree to take part in this study, you will complete questionnaires about symptoms you are having. You will be asked to fill these out 1 time a week during the first 2 months after surgery, 1 time a week during the first 3 months of a new therapy, and every 2 weeks at other times. The questionnaire will ask you to rate how severe your symptoms are and how the symptoms effect the activities of your daily life. The symptom questionnaire should take about 5 minutes to complete. You will complete the questionnaire during the first study visit and at your regular clinic visits.

Between clinic visits, you will be called every 1-2 weeks to complete the questionnaire using an automated telephone system. You can decide what time is most convenient for the automated phone system to call you. If you are not available when the automated system calls, it will call you again at a later time. If you are not reached by the automated phone system after several tries, the study staff will call you. You will be given a secure user name and identification number to use with the automated phone system. The study staff will teach you how to use the automated phone system.

At the clinic visit closest to 3 months after you start the study, you may be seen by a research staff member a second time 1 to 3 days after you completed the symptom questionnaire and asked to fill out the symptom questionnaire again. The research staff member may contact you by phone prior to this clinic visit to arrange times to meet you for the 2 assessments.

Quality-of-Life/Demographic Questionnaires:

At the first visit and the regular clinic visits, you will also rate your overall quality-of-life. This should take about 1 minute to complete.

At the first visit, you will also be asked some demographic questions (such as your age and marital status). Answering these questions should take about 1 minute.

Opinion Questionnaire:

If you are 1 of the first 40 patients enrolled in the study, you will be asked questions about your opinion of the symptom questionnaire at the clinic visit closest to 3 months after you start the study. For example, you will be asked if the symptom questionnaire was easy to understand and complete, and if there were any other questions that should be included. The study staff will use your opinion to decide if changes should be made to the questionnaire or if important symptom questions are missing from the questionnaire. This questionnaire should take about 5 minutes to complete.

Length of Study:

You will be on study for 1 year. You will be off study after you complete the last symptom questionnaire.

This is an investigational study.

Up to 188 participants will take part in this study. Up to 150 participants will be enrolled in Part 3 of this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older (Patient and family caregiver only)
2. Ability to speak and read English (All participants)
3. Residing where IVR service is available (Part 3, Patient only)
4. Diagnosis of GIST confirmed by pathological analysis (Patient only)
5. Starting new treatment (either surgical or medical) and planning to be followed at M.D. Anderson Cancer Center (Part 3, Patient only)
6. Written consent to participate (All participants)
7. At least 3 months from start of initial treatment (surgical or medical) for GIST (Part 2, Patient only)
8. Family caregiver also willing to receive packet for expert panel participation (Part 2, Patient only)
9. Physician or nurse with at least 5 years experience caring for patients with GIST (Professional expert only)
10. At least one publication in the last 5 years dealing with GIST (Physician professional expert only)
11. Identification as a family caregiver by a patient with GIST (Family caregiver only)
12. Patient also willing to receive packet for expert panel participation (Family caregiver only)

Exclusion Criteria:

1. Medical condition or impaired performance status that would preclude participation in the study (Patient only)
2. Diagnosis of active psychosis or severe cognitive impairment as determined by primary physician (Patient only)
3. Active treatment (systemic drug therapy or radiation therapy) for a second malignancy (Patient only)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: UT MD Anderson Cancer Center Sarcoma and Surgical Oncology Clinics GIST Patients, their caregivers, doctors and nurses who are 18 years or older.
Sampling Method: Non-Probability Sample
Enrollment: 187 (Actual)
Dates: Start 2010-07-29 (Actual); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Questionnaire Responses to Symptom Inventory for Gastrointestinal Stromal Tumors | Patients will be followed on study for 1 year regardless of changes in disease stage or treatments.
  Descriptive statistics used to assess the distributional characteristics and demographics of the study population and to report how patients rate symptom severity and interference with function.

CONTACTS AND LOCATIONS:
Overall Officials: Loretta A. Williams, PhD, MSN, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org